CLINICAL TRIAL: NCT07158242
Title: A Phase III Randomized Double-Blind Multi-Center Treat-Through Study to Evaluate the Pharmacokinetics, Safety and Efficacy of Induction and Maintenance Therapy With Afimkibart (RO7790121) in Children Aged 2 - 17 Years With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety and Efficacy of Afimkibart (RO7790121) in Children With Moderately to Severely Active Ulcerative Colitis
Acronym: AMETRINE-PEDS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA45905; 2025-522518-22-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Moderately to Severely Active Ulcerative Colitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Afimkibart Dose A (Experimental): Participants will receive Afimkibart intravenously (IV) followed by Afimkibart subcutaneous (SC) injection.
  Interventions: Drug: Afimkibart
- Afimkibart Dose B (Experimental): Participants will receive Afimkibart IV followed by Afimkibart SC.
  Interventions: Drug: Afimkibart

INTERVENTIONS:
Drug: Afimkibart — Afimkibart will be administered as IV infusion. Afimkibart will be administered as SC injection.
  Other Names: PF-06480605; RVT-3101; RG6631; RO7790121

SUMMARY:
This Phase III, randomized, double-blind, multicenter, induction and maintenance study will evaluate the safety and efficacy of Afimkibart (RO7790121) in pediatric participants with moderate to severe active ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Bodyweight >= 10 kilogram (kg)
* Confirmed diagnosis of UC
* Demonstrated intolerance or inadequate response (IR) to one or more of the following categories of drugs: systemic corticosteroids, immunomodulators, and/or biologic therapies as outlined in the protocol

Exclusion Criteria:

* Monogenic disorder pertaining to infant onset inflammatory bowel disease (IBD)
* Current diagnosis of Crohn's disease (CD), abdominal/intrabdominal/perianal fistula and/or abscess, indeterminant colitis, IBD-unclassified, microscopic colitis, ischemic colitis, infectious colitis, radiation colitis, or active diverticular disease
* Presence of an ostomy or ileoanal pouch
* Current diagnosis or suspicion of primary sclerosing cholangitis
* Any major surgery within 6 weeks prior to screening or a major planned surgery during the study
* Active tuberculosis (TB) infection suggested by positive TB testing, clinical symptoms, and/or chest imaging (X-ray or CT)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Remission at Week 12 | At Week 12
Percentage of Participants with Clinical Remission at Week 52 | At Week 52

SECONDARY OUTCOMES:
Change from Baseline in Pediatric Ulcerative Colitis Activity Index (PUCAI) Response | From Baseline, at Week 12
Percentage of Participants with PUCAI Remission | At Week 12
Change from Baseline in Tummy Ulcerative Colitis (TUMMY-UC) Scores | From Baseline to Week 12
Percentage of Participants with Endoscopic Improvement | At Week 12
Percentage of Participants with Histologic Improvement | At Week 12
Percentage of Participants with Histologic-endoscopic Mucosal Improvement | At Week 12
Percentage of Participants with Histologic-endoscopic Mucosal Remission | At Week 12
Change from Baseline in PUCAI Response at Week 52 | From Baseline, at Week 52
Percentage of Participants with PUCAI Remission at Week 52 | At Week 52
Change from Baseline in TUMMY-UC Scores | From Baseline to Week 52
Percentage of Participants with Endoscopic Improvement | At Week 52
Percentage of Participants with Histologic Improvement | At Week 52
Percentage of Participants with Histologic-endoscopic Mucosal Improvement | At Week 52
Percentage of Participants with Histologic-endoscopic Mucosal Remission | At Week 52
Percentage of Participants with Clinical Remission without the use of Corticosteriods | At Week 52
Percetage of Participants with Adverse Events (AEs) | From Baseline up to approximately 4 years
Serum Concentartion of Afimkibart | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing